CLINICAL TRIAL: NCT07396077
Title: Multimodal Physiological Reserve Optimizing Prehabilitation Program (PHYSIO-Prehab) in the Chinese Elderly With Spine Surgery
Brief Title: Pre-operative Risk Assessment Combined With Targeted Intervention in the Chinese Elderly With Spine Surgery II
Acronym: PRACTICE-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Xuanwu_PRACTICE-2
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Spine Degeneration; Lumbar Degenerative Disease; Frail Elderly; Enhanced Recovery After Surgery (ERAS) Protocol; Prehabilitation
Keywords: Prehabilitation; ERAS; lumbar fusion; ADL

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHYSIO-Prehab group (Experimental): The intervention group will receive a 6-week PHYSIO-Prehab multimodal prehabilitation program care. It includes 3 biweekly supervised group sessions and home-based multicomponent exercise. Additional interventions cover nutritional optimization, comorbidity management (targeting anemia, hypertension, and diabetes), and cognitive prehabilitation with brain protection measures.
  Both groups will receive consistent perioperative ERAS care implemented by the orthopedic department since January 2019, including multimodal and preemptive analgesia, inspiratory muscle training, minimal intravenous fluid administration, early urinary tube removal, avoidance of mechanical bowel preparation, no prolonged fasting, and antithrombotic prophylaxis
  Interventions: Other: Multimodal physiological reserve optimizing prehabilitation program
- Usual care group (Active Comparator): Participants in the group will receive standard care per the enhanced recovery protocol for lumbar fusion in older adults, including pre-admission health education on smoking/excessive drinking cessation, optimization of severe comorbidities, and general nutritional education.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Multimodal physiological reserve optimizing prehabilitation program — The PHYSIO-Prehab program features targeted multimodality integration, addressing the unmet need for surgery-specific preoperative interventions in elderly lumbar fusion patients. Its innovations lie in three aspects: first, it combines supervised group sessions with home-based exercise, balancing professional guidance and practical feasibility, and adjusts intensity via the Borg 10-point scale to fit individual tolerance. Second, it goes beyond conventional prehabilitation by integrating nutritional optimization, comorbidity management and cognitive prehabilitation, targeting physiological reserve deficits and frailty-related risks. Third, it is tailored to lumbar spinal disease characteristics, optimizing exercise modalities to avoid lumbar burden, which overcomes the limitations of general frailty interventions and enhances relevance to surgical recovery needs.
  Arms: PHYSIO-Prehab group
Other: Usual Care — Both groups will receive consistent perioperative ERAS care implemented by the orthopedic department since January 2019, including multimodal and preemptive analgesia, inspiratory muscle training, minimal intravenous fluid administration, early urinary tube removal, avoidance of mechanical bowel preparation, no prolonged fasting, and antithrombotic prophylaxis.
  Arms: Usual care group

SUMMARY:
This multicenter, parallel-group, assessor-blinded randomized controlled trial will enroll 248 adults aged ≥75 years with degenerative lumbar spinal diseases scheduled for elective lumbar fusion surgery, and they will be randomized 1:1 into the intervention and usual care groups. The intervention group will receive a 6-week PHYSIO-Prehab multimodal prehabilitation program, including multicomponent exercise, nutritional intervention, comorbidity optimization, and cognitive prehabilitation with brain protection strategies. The control group will receive standard health education provided via a manual, and both groups will receive consistent perioperative Enhanced Recovery After Surgery care. The primary outcome will be the change in Barthel Index (a tool for assessing independence in activities of daily living) from baseline to 30 days postoperatively; secondary outcomes will include pain scores, disability, patient satisfaction, and the 30-day postoperative Comprehensive Complication Index. The trial will initiate recruitment in April 2026 and conclude in December 2027, aiming to evaluate the feasibility and efficacy of PHYSIO-Prehab and provide high-quality evidence for patient-centered perioperative care pathways in this population.

DETAILED DESCRIPTION:
Degenerative lumbar spinal diseases are a leading cause of pain, disability, and reduced quality of life among older adults. As the global population ages rapidly, the volume of elderly patients undergoing elective lumbar fusion surgery will rise significantly. However, this cohort will face elevated risks of postoperative complications and delayed recovery of independence in activities of daily living, due to age-related decline in physiological reserve and multiple comorbidities. Enhanced Recovery After Surgery programs have shown value in reducing complications and accelerating recovery, but most focus on intraoperative and postoperative care, lacking targeted preoperative interventions for older adults with frailty or impaired physical function. Prehabilitation, a proactive preoperative strategy to enhance functional capacity and resilience to surgical stress, holds potential for improving postoperative outcomes, yet high-quality randomized trials in lumbar spinal surgery remain scarce. The PRACTICE-2 trial will address this evidence gap by evaluating a tailored multimodal prehabilitation program (PHYSIO-Prehab) for this specific population.

This multicenter, parallel-group, assessor-blinded randomized controlled trial will enroll 248 adults aged ≥75 years with degenerative lumbar spinal diseases who are scheduled for elective lumbar fusion surgery. Eligible patients will be randomized at a 1:1 ratio into the intervention group and the usual care group via stratified block randomization, with stratification by frailty status (frail vs. prefrail/non-frail) and participating center to balance key prognostic factors. The intervention group will receive a 6-week PHYSIO-Prehab program, consisting of 3 biweekly supervised group sessions (90 minutes each, including 60 minutes of lectures and 30 minutes of group discussion), plus home-based multicomponent exercise (resistance, balance, aerobic, and stretching training; 3 non-consecutive full sessions per week, with low-intensity walking on other days, adjusted based on the Borg 10-point scale). Additional interventions will include nutritional optimization (based on Mini Nutritional Assessment scores), comorbidity management (targeting anemia, hypertension, and diabetes), and cognitive prehabilitation with brain protection measures. The control group will receive standard health education provided via a manual, and both groups will receive consistent perioperative Enhanced Recovery After Surgery care as implemented by the participating hospitals.

The primary efficacy outcome will be the change in Barthel Index of Activities of Daily Living (0-20 points, with higher scores indicating better independence in basic daily activities such as feeding, dressing, and mobility) from baseline to 30 days postoperatively. Secondary efficacy outcomes will include the proportion of patients achieving full independence in activities of daily living (Barthel Index of Activities of Daily Living = 20) at 30 days postoperatively, Numeric Rating Scale scores for back and leg pain, Oswestry Disability Index, and patient satisfaction assessed via the 4-point North American Spine Society scale. The primary safety outcome will be the occurrence of severe or multiple complications, defined as a Comprehensive Complication Index greater than 20 within 30 days postoperatively. Secondary safety outcomes will include primary and total hospital length of stay, non-home discharge, and unplanned readmissions within 30 days postoperatively. The trial will initiate recruitment in April 2026, conclude in December 2027, and use R software for statistical analysis under a modified intention-to-treat principle, aiming to provide high-quality evidence for optimizing patient-centered perioperative care pathways for older adults undergoing lumbar fusion surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥75 years at the time of screening
2. Voluntarily sign the informed consent form
3. Clinically diagnosed with degenerative lumbar spinal disorders with duration of symptoms >6 months
4. Requiring elective lumbar fusion surgery (single-level or multi-level, open or minimally invasive approach)
5. No severe cognitive impairment (Mini-Mental State Examination score > 9)
6. Scheduled to undergo surgery within 6-8 weeks after screening (allowing completion of the 6-week prehabilitation program)

Exclusion Criteria:

1. Scheduled to undergo other emergency surgery or day surgery
2. Urgent medical conditions requiring priority management before spinal surgery
3. With spinal disorders other than degenerative diseases (spinal fracture, tumor, metastasis, infection, ankylosing spondylitis, scoliosis with Cobb angle >40°)
4. With contraindications to prehabilitation exercise (New York Heart Association Class IV heart failure, unstable angina, uncontrolled hypertension [systolic BP ≥180 mmHg or diastolic BP ≥110 mmHg despite medication])
5. With severe functional disability for other disorders or long-term bedridden status unable to perform basic physical activities
6. With allergy or intolerance to nutritional supplements used in the prehabilitation program
7. Participating in another clinical trial involving prehabilitation, perioperative intervention, or spinal surgery within 3 months before screening

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2026-04-25 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Barthel ADL Index from baseline to 30 days postoperatively | Within 30 days after surgery
  Primary efficacy outcome
30-day postoperative Comprehensive Complication Index | Within 30 days after surgery
  The proportion of participants with a Comprehensive Complication Index > 20

SECONDARY OUTCOMES:
30-day Barthel ADL Index postoperatively | Within 30 days after surgery
30-day postoperative Comprehensive Complication Index | Within 30 days after surgery
Length of hospital stay | Within 30 days after surgery
  Primary and total length of hospital stay
NRS for back and leg pain on day 30 after surgery | Within 30 days after surgery
North American Spine Society scale of satisfaction on day 30 after surgery | Within 30 days after surgery
Oswestry Disability Index on day 30 after surgery | Within 30 days after surgery
30-day non-home discharge postoperatively | Within 30 days after surgery
30-day unplanned readdmission postoperatively | Within 30 days after surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillis C, Ljungqvist O, Carli F. Prehabilitation, enhanced recovery after surgery, or both? A narrative review. Br J Anaesth. 2022 Mar;128(3):434-448. doi: 10.1016/j.bja.2021.12.007. Epub 2022 Jan 7. PMID 35012741
- [Background] Debono B, Wainwright TW, Wang MY, Sigmundsson FG, Yang MMH, Smid-Nanninga H, Bonnal A, Le Huec JC, Fawcett WJ, Ljungqvist O, Lonjon G, de Boer HD. Consensus statement for perioperative care in lumbar spinal fusion: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Spine J. 2021 May;21(5):729-752. doi: 10.1016/j.spinee.2021.01.001. Epub 2021 Jan 12. PMID 33444664
- [Background] Veronesi F, Borsari V, Martini L, Visani A, Gasbarrini A, Brodano GB, Fini M. The Impact of Frailty on Spine Surgery: Systematic Review on 10 years Clinical Studies. Aging Dis. 2021 Apr 1;12(2):625-645. doi: 10.14336/AD.2020.0904. eCollection 2021 Apr. PMID 33815887
- [Background] O'Lynnger TM, Zuckerman SL, Morone PJ, Dewan MC, Vasquez-Castellanos RA, Cheng JS. Trends for Spine Surgery for the Elderly: Implications for Access to Healthcare in North America. Neurosurgery. 2015 Oct;77 Suppl 4:S136-41. doi: 10.1227/NEU.0000000000000945. PMID 26378351
- [Background] Katz JN, Zimmerman ZE, Mass H, Makhni MC. Diagnosis and Management of Lumbar Spinal Stenosis: A Review. JAMA. 2022 May 3;327(17):1688-1699. doi: 10.1001/jama.2022.5921. PMID 35503342